CLINICAL TRIAL: NCT01610778
Title: A Randomized, Double-blind, Cross-over Study to Assess Efficacy of 5-Aminolevulinic Acid in Type 2 Diabetic Patients on Medication.
Brief Title: Effects of 5-Aminolevulinic Acid on Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: SBI Pharmaceuticals Co, Ltd. (Industry)
Responsible Party: Principal Investigator, Fumiko Higashikawa, Associate professor, Hiroshima University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: eki-541
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Type 2 Diabetes on Medication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Supplement (Experimental)
  Interventions: Dietary Supplement: 5-aminolevulinic acid phosphate

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Placebo
Dietary Supplement: 5-aminolevulinic acid phosphate
  Arms: Supplement

SUMMARY:
This study is designed to evaluate efficacy of 5-aminolevulinic acid in subjects with type 2 diabetes on medication.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients on medication
* HbA1c ≤ 9.0% (as JDS values, which is equivalent to HbA1c ≤ 9.4% as NGSP values)
* On stable treatment of diabetes for at least the last 3 months
* With permission to attend the clinical trial from the primary doctor

Exclusion Criteria:

* On insulin therapy
* BMI ≤ 18 kg/m2 or ≥ 30 kg/m2
* History of porphyria, hemochromatosis, or viral hepatitis
* Pregnant or nursing a child
* Heart disease
* Renal or hepatic dysfunction
* Participation in any clinical trial within 90 days of the commencement of the trial

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Fasting glucose level | Every 4 weeks (Overall 36 weeks)
HbA1c level | Every 4 weeks (Overall 36 weeks)
Glycoalbumin level | Every 4 weeks (Overall 36 weeks)

SECONDARY OUTCOMES:
Fasting insulin level | Every 4 weeks (Overall 36 weeks)
1,5-AG level | Every 4 weeks (Overall 36 weeks)
Serum C-peptide level | Every 4 weeks (Overall 36 weeks)
HOMA-R | Every 4 weeks (Overall 36 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Hiroshima University, Hiroshima, Japan